CLINICAL TRIAL: NCT06185010
Title: Effects of Different Resistance Training Volumes on Cognitive Function, Oxidative Stress, Immunological Response, Lipid Profile, Glycemic Status, Liver Function, Muscle Function, Hemodynamic Response, and Physical Performance in Individuals With Mild Cognitive Impairment
Brief Title: Resistance Training to Individuals for Cognitive Impairment With Dementia
Acronym: TRAIN4BRAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beira Interior (Other)
Collaborators: Research Center in Sports Sciences, Health Sciences and Human Development (Other)
Responsible Party: Principal Investigator, Nuno Miguel Pintassilgo da Silva Fonseca, Researcher, University of Beira Interior
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: University of Beira Interior
Record Dates: First submitted 2023-12-14; First posted 2023-12-29 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Mild Cognitive Impairment; Mild Dementia
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- One Resistance Training Set (Single Session) (Experimental): The participants will perform one resistance training session with one set.
  Interventions: Other: One Resistance Training Set (Single Session)
- Three Resistance Training Sets (Single Session) (Experimental): The participants will perform one resistance training session with three sets.
  Interventions: Other: Three Resistance Training Sets (Single Session)
- One Resistance Training Set (8 Weeks) (Experimental): The participants will perform eight weeks of resistance training (two sessions per week, separated by 72 hours of rest) with one set.
  Interventions: Other: One Resistance Training Set (8 Weeks)
- Three Resistance Training Sets (8 Weeks) (Experimental): The participants will perform eight weeks of resistance training (two sessions per week, separated by 72 hours of rest) with three sets.
  Interventions: Other: Three Resistance Training Sets (8 Weeks)
- Control (8 Weeks) (Experimental): The participants will not perform any form of physical exercise during the intervention period of eight weeks.
  Interventions: Other: Control (8 Weeks)

INTERVENTIONS:
Other: One Resistance Training Set (Single Session) — The participants will perform a resistance training session with one set per exercise. The training sequence will be the following: i) 10 minutes of warm-up walking on the treadmill at 50% of maximal walking velocity, ii) 1 set of 10 repetitions at 60% of one-repetition maximum (1RM) in the leg press, iii) 1 set of 10 repetitions at 55% 1RM in the chest press, iv) 1 set of 10 repetitions in the sit-to-stand exercise, v) 1 set of 10 repetitions in the 1-kg medicine ball throw exercise, and vi) 5 minutes walking on the treadmill at 60% of maximal walking velocity.
  Arms: One Resistance Training Set (Single Session)
Other: Three Resistance Training Sets (Single Session) — The participants will perform a resistance training session with three sets per exercise. The training sequence will be the following: i) 10 minutes of warm-up walking on the treadmill at 50% of maximal walking velocity, ii) 3 sets of 10 repetitions at 60% of one-repetition maximum (1RM) in the leg press, iii) 3 sets of 10 repetitions at 55% 1RM in the chest press, iv) 3 sets of 10 repetitions in the sit-to-stand exercise, v) 3 sets of 10 repetitions in the 1-kg medicine ball throw exercise, and vi) 5 minutes walking on the treadmill at 60% of maximal walking velocity.
  Arms: Three Resistance Training Sets (Single Session)
Other: One Resistance Training Set (8 Weeks) — The participants will perform eight weeks of resistance training with one set per exercise. The training sequence will be the following: i) 10 minutes of warm-up walking on the treadmill at 50% of maximal walking velocity, ii) 1 set of 10 repetitions between 50-70% of one-repetition maximum (1RM) in the leg press, iii) 1 set of 10 repetitions between 40-60% 1RM in the chest press, iv) 1 set of 6-12 repetitions in the sit-to-stand exercise, v) 1 set of 6-12 repetitions in the 1-kg medicine ball throw exercise, and vi) 5 minutes walking on the treadmill at 60% of maximal walking velocity.
  Arms: One Resistance Training Set (8 Weeks)
Other: Three Resistance Training Sets (8 Weeks) — The participants will perform eight weeks of resistance training with three sets per exercise. The training sequence will be the following: i) 10 minutes of warm-up walking on the treadmill at 50% of maximal walking velocity, ii) 3 sets of 10 repetitions between 50-70% of one-repetition maximum (1RM) in the leg press, iii) 3 sets of 10 repetitions between 40-60% 1RM in the chest press, iv) 3 sets of 6-12 repetitions in the sit-to-stand exercise, v) 3 sets of 6-12 repetitions in the 1-kg medicine ball throw exercise, and vi) 5 minutes walking on the treadmill at 60% of maximal walking velocity.
  Arms: Three Resistance Training Sets (8 Weeks)
Other: Control (8 Weeks) — The participants in the control group will maintain their regular daily activities without performing any form of physical exercise.
  Arms: Control (8 Weeks)

SUMMARY:
This research project aims to analyze the effects of different resistance training volumes on cognitive function, oxidative stress, immunological response, lipid profile, glycemic status, liver function, muscle function, hemodynamic response, and physical performance in individuals with mild cognitive impairment. First the investigators will analyze the effects of a single resistance training session (acute effects) with one and three sets on hemodynamic and physical performance in individuals with mild cognitive impairment. After, the investigators will analyze the effects of an 8-week resistance training program with one or three sets on cognitive function, oxidative stress, immunological response, lipid profile, glycemic status, liver function, muscle function, hemodynamic response, and physical performance in individuals with mild cognitive impairment. The investigators hypothesize that a single resistance training session of one or three sets will increase the acute hemodynamic and physical performance stress in individuals with mild cognitive impairment, although with a higher magnitude in the session with three sets. Furthermore, we hypothesize that eight weeks of resistance training with one or three sets will induce similar improvements in cognitive function, oxidative stress, immunological response, lipid profile, glycemic status, liver function, muscle function, hemodynamic response, and physical performance in individuals with mild cognitive impairment.

DETAILED DESCRIPTION:
Following specific inclusion and exclusion criteria (see Eligibility Criteria), participants will be recruited from residential care facilities or day centers. For the acute effects study (cross-over study), participants will randomly perform two resistance training sessions separated by one week of rest: i) one session with one set and ii) another session of three sets. The intensity of the exercises, number of repetitions, type and order of exercises, movement velocity, and rest time between exercises will be the same in both groups. Before, immediately after, and 72 hours after the sessions, a battery of tests will be applied to evaluate the changes in blood pressure, heart rate, tympanic temperature, medicine ball throw distance, five-repetition sit-to-stand time, and handgrip strength. Afterward, participants will be randomly assigned into a one-set or three-set group to perform an eight-week resistance training intervention. As for the acute effects study, the prescription of the other acute training variables will be the same for both groups. A control group (without any form of physical exercise), recruited at the beginning of the research project, will also be part of the study. Before and after the intervention, a battery of tests will be applied to determine the training program's impact on cognitive function, oxidative stress, immunological response, lipid profile, glycemic status, liver function, muscle function, hemodynamic response, and physical performance in individuals with mild cognitive impairment.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of mild cognitive impairment
* SPPB score ≥ 3 points
* Willingness to participate in the interventions and collaborate with the research team
* Must be able to provide informed consent (oral or written)

Exclusion criteria:

* Severe dementia
* Severe comorbidity that negatively influences participation in the intervention
* Color blindness
* Fractures in the last three months

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure (SBP) | Change from baseline to 0 minutes and 72 hours after the sessions
  In the cross-over study (acute effects), the SBP will be assessed through a blood pressure device.
Handgrip strength (HGS) | Change from baseline to 0 minutes and 72 hours after the sessions
  In the cross-over study (acute effects), the HGS will be assessed through an analogic dynamometer.
Dementia Rating Scale-2 (DRS-2) | Change from baseline to week 8
  In the eight-week study, the DRS-2 questionnaire will be applied to analyze the overall level of cognitive function through five subscales: attention, initiation/perseveration, construction, conceptualization, and memory.
Brain-Derived Neurotrophic Factor (BDNF) | Change from baseline to week 8
  In the eight-week study, the BDNF protein levels will be analyzed through specific blood testing kits.
Short Physical Performance Battery (SPPB) | Change from baseline until week 8
  In the eight-week study, the SPPB will determine the overall level of functional performance through three tests: balance (feet side by side, semi tandem, tandem), 4-meter walking, and 5-repetition sit-to-stand.

SECONDARY OUTCOMES:
Diastolic blood pressure (DBP) | Change from baseline to 0 minutes and 72 hours after the sessions
  In the cross-over study (acute effects), the DBP will be assessed through a blood pressure device.
Heart rate (HR) | Change from baseline to 0 minutes and 72 hours after the sessions
  In the cross-over study (acute effects), the HR will be assessed through a blood pressure device.
Tympanic temperature (TT) | Change from baseline to 0 minutes and 72 hours after the sessions
  In the cross-over study (acute effects), the TT will be assessed through a tympanic thermometer.
Five-repetition sit-to-stand (5STS) | Change from baseline to 0 minutes and 72 hours after the sessions
  In the cross-over study (acute effects), the 5STS time will be recorded through a chronometer.
1-kg Medicine Ball Throw (MBT) | Change from baseline to 0 minutes and 72 hours after the sessions
  In the cross-over study (acute effects), the MBT distance will be recorded with a tape measure.
Inflammatory markers | Change from baseline to week 8
  In the eight-week study, inflammatory markers (IL-6, TNF-α, and IL-10) will be analyzed through specific blood testing kits.
Oxidative stress | Change from baseline to week 8
  In the eight-week study, oxidative stress markers (carbonylated proteins) will be analyzed through specific blood testing kits.
Lipid Profile | Change from baseline to week 8
  In the eight-week study, the lipid profile (LDL, HDL, total cholesterol, triglycerides) will be analyzed through specific blood testing kits.
HbA1c | Change from baseline to week 8
  In the eight-week study, the HbA1c will be analyzed through specific blood testing kits.
Muscle Damage | Change from baseline to week 8
  In the eight-week study, the muscle damage (creatine kinase, lactate dehydrogenase, aspartate aminotransferase, and alanine aminotransferase) will be analyzed through specific blood testing kits.
One-repetition maximum (1RM) | Change from baseline to week 8
  In the eight-week study, a progressive loading test until reaching the 1RM will be applied in the horizontal leg press and seated chest press machines.
Load-velocity profiles | Change from baseline to week 8
  In the eight-week study, the load-velocity profiles will be analyzed using the velocity values (recorded with a linear velocity transducer) associated with the absolute loads used during the progressive loading tests in the horizontal leg press and seated chest press machines.
Ten-meters walking | Change from baseline to week 8
  In the eight-week study, the 10-meter walking time will be measured through a chronometer.
1-kg Medicine Ball Throw (MBT) | Change from baseline to week 8
  In the eight-week study, the MBT distance will be recorded with a tape measure.
Handgrip strength (HGS) | Change from baseline to week 8
  In the eight-week study, the HGS will be assessed through an analogic dynamometer.
6-Minute Walk Test (6MWT) | Change from baseline to week 8
  In the eight-week study, the 6MWT distance will be assessed by multiplying the number of total laps by the lap distance (e.g., 10 laps x 10 meters).

CONTACTS AND LOCATIONS:
Overall Officials: Mário C Marques, PhD, Principal Investigator — University of Beira Interior; Dulce Esteves, PhD, Principal Investigator — University of Beira Interior; Mikel Izquierdo, PhD, Principal Investigator — Universidad Pública de Navarra
Locations (1):
- University of Beira Interior, Covilha, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fonseca N, Esteves D, Marques DL, Fail LB, Sousa T, Pinto MP, Neiva HP, Izquierdo M, Marques MC. Acute and time-course changes in hemodynamic and physical performance parameters following single and multiple resistance training sets in cognitively impaired individuals: A randomized crossover study. Exp Gerontol. 2025 Mar;201:112688. doi: 10.1016/j.exger.2025.112688. Epub 2025 Jan 23. PMID 39854950